

Effects of time of day and menstrual cycle phase (low and high progesterone) on female's cognitive and strength performance.

NTC number: Approved: 05/01/2026



## **Consent Form**

**Study Title:** Effects of time of day and menstrual cycle phase (low and high progesterone) on female's cognitive and strength performance.

We are asking if you would like to take part in a research project that aims to investigate how time-of-day and levels of progesterone (a hormone which varies through the menstrual cycle) affect female's executive function (part of cognitive abilities) and muscle strength. The results of this study will reveal whether executive function and muscle strength fluctuate with time of day and menstrual cycle.

Before you consent to participating in the study, we ask that you read the participant information sheet and mark each box below with your initials if you agree. If you have any questions or queries before signing the consent form, please speak to the researcher Anna Stone.

| Name | of ResearcherDateDate |
|---|---|
| Name | of ParticipantDate |
| 8. | I consent to take part in the above study. |
| 7. | I understand that any information I give will remain confidential and anonymous unless it is thought that there is a risk of harm to myself or others, in which case the researcher may need to share this information with their research supervisor. |
| 6. | I consent to Lancaster University keeping the anonymised data for a period of 10 years after the study has finished, and for the fully anonymised research data to be stored indefinitely on the Open Science Framework. |
| 5. | I understand that the researcher will discuss data with their supervisor as needed. |
| 4. | I understand that once my data has been anonymised it might not be possible for it to be withdrawn, as such I have up until the end of my participation in the study to inform the researcher if I wish for my data to be withdrawn. |
| 3. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. |
| 2. | I confirm that I have had the opportunity to ask any questions and to have them answered. |
| 1. | I confirm that I have read the information sheet and fully understand what is expected of me within this study. |